CLINICAL TRIAL: NCT00380328
Title: An Open-label, Randomized, 2-period Crossover, Drug Interaction Study to Evaluate the Potential Pharmacokinetic Interaction Between Multiple Doses of Ketoconazole and a Single Dose of HKI-272 Administered Orally to Healthy Subjects
Brief Title: HKI-272 Ketoconazole Drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3144A1-106
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Pharmacokinetic; healthy subjects
MeSH Terms: interventions — neratinib

INTERVENTIONS:
Drug: neratinib — HKI-272

SUMMARY:
To investigate a potential pharmacokinetic drug interaction between HKI-272 and ketoconazole when co-administered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead ECG.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-10; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics; safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology